CLINICAL TRIAL: NCT03226509
Title: Transforming the Cascade of Hepatitis C Care
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Norman Randall Kolb, Principle Investigator; Associate Program Director UPMC Shadyside Family Medicine Residency, University of Pittsburgh
Other Study IDs: PRO16040427
Record Dates: First submitted 2017-02-27; First posted 2017-07-21 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C, Chronic
Keywords: cascade of care
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several factors are barriers to effective Hepatitis C care: 1) The majority of Hepatitis C Virus (HCV)-positive patients (45-85 percent) are unaware that they are infected; 2) Only a small minority of those in need of treatment receive it; 3) Members of minorities and older patients are even less likely to receive needed care; and 4) Until recently, even those who were treated had a low chance of clearing the virus or achieving cure; 5) It is possible that older attitudes and expectation of futility might continue to persist among patients and provider in primary care settings.

Community Health Centers are often the most culturally appropriate and accessible choices, particularly for underserved populations, with the benefit of ongoing trust and relationships with patients. Therefore, these can be ideal places to deliver complex HCV care if they possess the needed expertise. However, most community-based primary care and community health centers lack access to Hepatitis C evaluation and treatment services, leading to a major public health problem.

Thus, investigators propose to implement and evaluate a pragmatic trial to implement and evaluate a multi-disciplinary model for HCV treatment at Currently, the treatment initiation rates at each of these sites is estimated as less than 10%. The investigators hypothesize that our project will increase the rate of participation in all the steps of the HCV care cascade and ultimately lead to more than doubled rates of treatment uptake

DETAILED DESCRIPTION:
Primary Objective:

Determine uptake, effectiveness and safety of IFN-free, DAAs among "real world" patients, including those with multiple comorbidities, in the primary care setting.

Secondary Objective(s):

1. Demonstrate the transformation of the cascade of Hepatitis C Care at 3 primary care clinics in terms of changes from baseline in rates for rates of access to HCV care including HCV screening, evaluation, treatment consideration, treatment uptake, completion, loss to follow-up, and treatment success rate.
2. Advance understanding of hepatitis C related decision-making in the era of Interferon (IFN)-free Direct acting agents (DAAs) by examining the context, needs, motivators, barriers, and preferences among patients and providers to the delivery of hepatitis C treatment at primary care clinics

ELIGIBILITY:
Inclusion Criteria:

* All patients with detectable HCV RNA level, currently receiving care at any of these three community health centers

Exclusion Criteria:

* Criteria for automatic specialty referral (exclusion from treatment at community health centers) Child Turcotte Pugh Class B or C Any history of decompensated liver disease or hepatocellular carcinoma Evidence of renal disease (GFR <50) or coexisting autoimmune condition HIV of hepatitis B co-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with detectable HCV RNA level, currently receiving care at any of these three community health centers
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving sustained viral response 12 weeks post treatment (SVR 12) over a three year intervention period. | three years
  measure percentage of patients moving through the cascade of care to cure of condition (SVR 12)

SECONDARY OUTCOMES:
Rates of Hepatitis C Virus (HCV) screening | three years
  Percentage of at risk patients in the practice who have a completed HCV antibody test
Rate of Chronic Hepatitis C evaluation | three years
  Percentage of patients with a positive HCV antibody test who have a HCV polymerase chain reaction (PCR) viral load completed
Rate of treatment consideration | three years
  Percentage of consented patients with a positive HCV viral load who have a clinical evaluation and assessment of psychosocial readiness for treatment documented in the medical record
Rate of treatment uptake | three years
  Percentage of patients recommended for treatment who begin medical treatment
Rate of treatment completion | three years
  Percentage of patients that began treatment who complete the recommended course of therapy
Rate of patients lost to follow up | three years
  Percent of consented patients with a positive HCV viral load who are lost to follow up
Hepatitis C capacity building among family medicine physicians (provider practice and perceived confidence): | three years
  Endpoints related to HCV capacity building among family medicine physicians: Evaluate comfort and skill among family physicians to evaluate and treat HCV infection as measured on a qualitative survey of physicians

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Shadyside Family Health Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No